CLINICAL TRIAL: NCT06204367
Title: Evaluation of Lung Ultrasonography Findings in Newborns With Respiratory Syncytial Virus Bronchiolitis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Sevde Nur Vural, Asistant Doctor, Kırıkkale University
Other Study IDs: Kırıkkale Neonatology
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: RSV Infection; Bronchiolitis
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Bronchiolitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung Ultrasonografisi — It is aimed to compare the agreement between lung ultrasonography and clinical score in the diagnosis and follow-up of newborn babies who are followed up in the neonatal intensive care unit due to bronchiolitis caused by frequently encountered RSV and other viral factors.

SUMMARY:
Respiratory Syncytial Virus (RSV) is a seasonal, highly contagious pathogen belonging to the Pneumoviridae (genus orthopneumovirus), a family of negative-strand RNA viruses. Lung ultrasonography; Today, it has become frequently used in neonatal intensive care units because it is a diagnostic, useful, harmless, radiation-free, bedside, reproducible and practical method. The primary purpose of the study is to record lung ultrasound findings and score and thus to compare the agreement between lung ultrasonography and clinical score in the diagnosis and follow-up of newborn babies who are followed up in the neonatal intensive care unit due to bronchiolitis caused by RSV and other viral factors, which are frequently encountered.

DETAILED DESCRIPTION:
Respiratory Syncytial Virus (RSV) is a type of negative-strand RNA viruses. It is a seasonal, highly contagious pathogen belonging to the family Pneumoviridae (genus orthopneumovirus). RSV is a common cause of respiratory disease throughout life but is associated with significant morbidity and mortality, especially in infants and older adults.

RSV infections account for approximately 60% to 80% of bronchiolitis in infancy and 40% of pediatric pneumonias.

Bronchiolitis is an acute lower respiratory tract infection that affects children under one or two years of age and is the most common cause of hospitalization, according to American Academy of Pediatrics (AAP) guidelines. Diagnostic criteria for bronchiolitis are based on clinical history and examination.

Lung ultrasonography (LUS) was first used in adults in 1995, and in the last decade, lung ultrasound has proven to be a useful diagnostic tool in many pediatric and neonatal diseases, and its application and benefit in the treatment of bronchiolitis has been reported. Since AUS allows bedside assessment of the subpleural lung for density, thus reducing the quantitative ratio of airspace and space, it is reasonable to expect that a combination of clinical and ultrasound parameters may be useful. Studies have shown that qualitative and quantitative lung ultrasound findings suggest a relationship with the severity of bronchiolitis and are useful in the follow-up of patients.

Caiulo et al. They showed that AUS is a valuable tool in the diagnosis of bronchiolitis.

However, data on lung ultrasound in newborns with viral lower respiratory tract infections are quite limited.

Lung ultrasonography; Today, it has become frequently used in neonatal intensive care units because it is a diagnostic, useful, harmless, radiation-free, bedside, reproducible and practical method. In our clinic, lung ultrasonography is performed on babies hospitalized with respiratory distress. Images will be obtained using the linear probe of the device to be used for AUS. Brat et al. AUS scoring specified in the studies of Raimondi et al. and Raimondi et al. will be used.

Accordingly, both lungs will be evaluated as three areas on the right and left (anterior upper, anterior lower and lateral) and will be scored separately. Parasternal with anterior axillary line in front The area between the line is divided into two by the line passing from the nipple. The upper part is considered as the upper anterior region and the lower part is considered as the lower anterior region. The area in the middle of the anterior and posterior axillary lines is called the lateral region.

is evaluated. Each field is given a score of 0 to 3. If there were A lines, 0 points were given. If there were more than 3 B lines in an area, 1 point was given. If the B lines were very dense and there was no A line, it was evaluated as white lung and 2 points were given. If there was a consolidation image in AUS, 3 points were given. The total score was evaluated as a maximum of 18. In this study, newborn babies who were admitted and admitted to the Neonatal Intensive Care Unit of Kırıkkale University Faculty of Medicine Hospital with symptoms of viral lower respiratory tract diseases between 18/12/2023 and 01/06/2023 were clinically diagnosed with 40% of their O2 need at the 24th hour of hospitalization. Lung ultrasonography was planned to be performed in cases where the patient was overweight and/or required pressure or was intubated, and at the time of discharge. Demographic characteristics, symptoms, all routine laboratory and radiological imaging of newborn babies, and additional pathogen or pathogens will be obtained from the file information. The parameters to be recorded are shown in the Case Report Form. The primary purpose of the study is to record lung ultrasound findings and score and thus to compare the agreement between lung ultrasonography and clinical score in the diagnosis and follow-up of newborn babies who are followed up in the neonatal intensive care unit due to bronchiolitis caused by RSV and other viral factors, which are frequently encountered.

ELIGIBILITY:
Inclusion Criteria:

* All newborns hospitalized with viral lower respiratory tract findings in the neonatal intensive care unit of Kırıkkale University Faculty of Medicine Hospital
* Patients with study approval
* Patients who underwent lung ultrasonography were included in the study.

Exclusion Criteria:

* Newborns who do not lie down due to viral lower respiratory tract infection
* Patients without study consent
* Patients for whom lung ultrasonography could not be performed

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborn
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Lung ultrasonography | 5 months
  It is aimed to compare the agreement between lung ultrasonography and clinical score in the diagnosis and follow-up of newborn babies who are followed up in the neonatal intensive care unit due to bronchiolitis caused by frequently encountered RSV and other viral factors.

SECONDARY OUTCOMES:
lung radrology | 5 months
  The aim of using lung ultrasound in the clinical follow-up of newborn babies diagnosed with bronchiolitis caused by respiratory viral factors is to reduce the number of lung films and therefore reduce radiation exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Sevde Nur nu Vural, Asistant Dr, Study Chair — KIRIKKALE UNİVERSİTY FACULTY OF MEDİCİNE
Locations (1):
- Kırıkkale University Faculty of Medicine, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Azzari C, Baraldi E, Bonanni P, Bozzola E, Coscia A, Lanari M, Manzoni P, Mazzone T, Sandri F, Checcucci Lisi G, Parisi S, Piacentini G, Mosca F. Epidemiology and prevention of respiratory syncytial virus infections in children in Italy. Ital J Pediatr. 2021 Oct 2;47(1):198. doi: 10.1186/s13052-021-01148-8. PMID 34600591
- [Background] Demont C, Petrica N, Bardoulat I, Duret S, Watier L, Chosidow A, Lorrot M, Kieffer A, Lemaitre M. Economic and disease burden of RSV-associated hospitalizations in young children in France, from 2010 through 2018. BMC Infect Dis. 2021 Aug 2;21(1):730. doi: 10.1186/s12879-021-06399-8. PMID 34340679
- [Background] American Academy of Pediatrics Committee on Infectious Diseases; American Academy of Pediatrics Bronchiolitis Guidelines Committee. Updated guidance for palivizumab prophylaxis among infants and young children at increased risk of hospitalization for respiratory syncytial virus infection. Pediatrics. 2014 Aug;134(2):415-20. doi: 10.1542/peds.2014-1665. PMID 25070315
- [Background] Nair H, Nokes DJ, Gessner BD, Dherani M, Madhi SA, Singleton RJ, O'Brien KL, Roca A, Wright PF, Bruce N, Chandran A, Theodoratou E, Sutanto A, Sedyaningsih ER, Ngama M, Munywoki PK, Kartasasmita C, Simoes EA, Rudan I, Weber MW, Campbell H. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. Lancet. 2010 May 1;375(9725):1545-55. doi: 10.1016/S0140-6736(10)60206-1. PMID 20399493
- [Background] Brat R, Yousef N, Klifa R, Reynaud S, Shankar Aguilera S, De Luca D. Lung Ultrasonography Score to Evaluate Oxygenation and Surfactant Need in Neonates Treated With Continuous Positive Airway Pressure. JAMA Pediatr. 2015 Aug;169(8):e151797. doi: 10.1001/jamapediatrics.2015.1797. Epub 2015 Aug 3. PMID 26237465
- [Derived] Tandircioglu UA, Koral U, Menemen SN, Alan S. Comparison of clinical findings and lung ultrasound scores in newborns with RSV and non-RSV viral lower respiratory tract infections: a prospective observational study. Eur J Pediatr. 2025 Dec 11;185(1):6. doi: 10.1007/s00431-025-06687-4. PMID 41379208